CLINICAL TRIAL: NCT04467710
Title: Treatment of Common Bile Duct Stones in a Laparoscopic Center : What Are the Limits and When Should we Call the Endoscopist ? Observationnal Study Between 2007-2019
Brief Title: Laparoscopic Treatment of Common Bile Duct Stones : What Are the Limits and When Should we Call the Endoscopist ?
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0001
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-07

CONDITIONS: Laparoscopic; Common Bile Duct Stone With Chronic Cholecystitis
Keywords: Common bile duct stones; Laparoscopic common bile duct exploration (LCBDE); ERCP; Morbimortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Success of LCBDE: Patients with a fully laparoscopic surgical treatment of common bile duct stones
  Interventions: Procedure: Laparoscopic common bile duct exploration.
- Failure of LCBDE: Patients with a laparoscopic cholecystectomy but an endoscopic treatment of common bile duct stone with an ERCP performed intra, per or postoperatively
  Interventions: Procedure: Laparoscopic common bile duct exploration.

INTERVENTIONS:
Procedure: Laparoscopic common bile duct exploration. — Laparoscopic common bile duct exploration. ERCP (Endoscopic Retrograde Cholangiopancreatography) with sphincterotomy : : removal of common bile duct stones trought the cystic duct (transcystically) with a Dormia or a choledoscope, or throught the common bile duct with a choledoscope introduced throught an incision of the common bile duct.
  ERCP with sphincterotomy: removal of common bile duct stones throught the duodenal papilla, and a sphincterotomy of the oddi sphincter during the same time.

SUMMARY:
The aim of this study was to identify some risk factors of failure of surgical management of common bile duct stones, in our center between 2007 and 2019.

DETAILED DESCRIPTION:
Lithiasis disease represents a real public health problem. Indeed, 10% of the general population is asymptomatic carrier of gallbladder stones and among them, 35% will present a symptomatic form which will cause the indication of cholecystectomy. As a result, around 120,000 cholecystectomies are performed per year in France, and around 750,000 in the United States for this indication. Cholecystectomy is therefore the most widely performed procedure in the world. However, in 3 to 20% of cases, common bile duct stones will be associated and to be treated. Different strategies are proposed: a treatment called "all surgical" or an endoscopic treatment (usually a sphincterotomy) before, after or during a cholecystectomy. The investigators defined two groups of patients: one group with success of fully laparoscopic surgical treatment (cholecystectomy and laparoscopic exploration of the common bile duct at the same time), and one group treated by laparoscopic cholecystectomy and management of the common bile duct stone(s) by an ERCP performed intra, per ou postoperatively. The primary outcome was the failure of surgical management, defined as the requirement of ERCP for extraction of common bile duct stones, which permit us to identify risk factors of failure in the fullfil surgical treatment process. The secondary outcome was to study the morbimortality in each group, and length of stay.

ELIGIBILITY:
Inclusion criteria:

* More than 18 years old
* Between 2007 and 2019
* Montpellier University Hospital
* Laparoscopic cholecystectomy for symptomatic cholelithiasis associated to common bile duct stones
* Common bile duct stones highlighted on preoperative imaging or intraoperative cholangiography
* Common bile duct stones treated during the same hospital stay surgically or endocopically

Exclusion criteria:

* Laparotomy
* Previous ERCP
* Less than 18 years old
* Lost to follow up
* Lack of data > 10%
* Other surgical procedure associated at the same time
* Previous cholecystectomy
* Caroli's disease
* Severe cholangitis or acute pancreatitis
* Pigmentary or hydatic lithiasis
* Laparoscopic cholecystectomy for other indication than symptomatic cholelithiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged more than 18, hospitalized in Montpellier University Hospital between 2007 and 2019 requiring a laparoscopic cholecystectomy for symptomatic biliary disease associated to a common bile duct stone highlighted on preoperative imaging or intraoperative cholangiography, which will be treated surgically or endoscopically during the same hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
morbimortality | 1 day
  Clavien dindo classification

SECONDARY OUTCOMES:
risk factors of total laprascopic treatment failure. | 1 day
  risk factors of total laprascopic treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid HERRERO, MD, PHD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Genet D, Souche R, Roucaute S, Borie F, Millat B, Valats JC, Fabre JM, Herrero A. Upfront Laparoscopic Management of Common Bile Duct Stones: What Are the Risk Factors of Failure? J Gastrointest Surg. 2023 Sep;27(9):1846-1854. doi: 10.1007/s11605-023-05687-9. Epub 2023 Apr 27. PMID 37106206